CLINICAL TRIAL: NCT01142297
Title: A Randomized, Controlled Trial Comparing the Stability of SLA Implants and SLActive Implants Using Resonance Frequency Analysis for Patients With Type 2 Diabetes Mellitus
Brief Title: Comparative Study of Implant Surfaces to Enhance Stabilization in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0156H
Record Dates: First submitted 2010-04-29; First posted 2010-06-11 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2016-09

CONDITIONS: Partially Edentulous Mandible; Type 2 Diabetes
Keywords: dental implant; implant stabilization; type 2 diabetes; glycated hemoglobin 8.0-12.0%
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dental implant (Other): standard SLA surface and chemically modified surface
  Interventions: Device: dental implant and modified dental implant

INTERVENTIONS:
Device: dental implant and modified dental implant — standard SLA surface and chemically modified surface

SUMMARY:
This study compares the patterns of dental implant stabilization between a standard and chemically modified implant surface in patients with type 2 diabetes. It is hypothesized that the chemically modified surface will enhance early healing events (first 4 months following placement)in diabetes patients with compromises in rate of implant integration.

DETAILED DESCRIPTION:
This is a prospective randomized study design whereby type 2 diabetic patients will receive 2 implants in the mandible or maxilla to assess implant integration. One implant will be a regular SLA implant; the other will have a SLActive surface. The primary objective of this randomized controlled study is to evaluate the stability of Straumann 4.1 mm diameter implants in the posterior mandible or maxilla of type 2 diabetic patients during the first 12 weeks after implantation using resonance frequency analysis. The control implant is a standard Straumann implant with an SLA® surface and the test implant the same implant design with SLActive® surface. Assessments will utilize resonance frequency analysis (RFA), as a measure of implant integration, and clinical outcomes of implant success. This study will enroll type 2 diabetes patients having glycated hemoglobin (HbA1c) levels from 8.0% to 12% at baseline.

The primary objective is to test for statistically significant differences in ISQ values between the test and control implants at 2, 3, 4, 6, 7, 8 weeks and 3 months after surgery. If a difference of 2 Osstell RFA ISQ units is detected at any time point it will be considered that the implant having achieved the higher value is better osseointegrated. This split-mouth study design will assess changes in implant stability from baseline as the primary outcome at the implant level. This study will require 20 patients to detect this difference (SD=2.0 ISQ units) with a power of 80% at the P=0.05 level.

Secondary objectives include:

* Implant survival and implant success at 1-year post loading.
* The nature and frequency of adverse events/complications between the 2 groups will be compared.
* Prosthesis success

ELIGIBILITY:
Inclusion Criteria:

* Males and females must be at least 18 years of age, and having a diagnosis of type 2 diabetes mellitus occurring over 1 year prior to enrollment (self-reported and verified with physician report, test results, and/or treatment record)
* Type 2 diabetic patients may be on a modified diet, oral medication, insulin, or combination therapies
* Glycated hemoglobin A1c (HbA1c) levels of at least 8.0% up to and including 12.0% as reported within 4 weeks of implant placement
* Have at least two missing teeth in the posterior mandible in FDI positions 4, 5, 6, or 7
* The tooth at the implant site must have been extracted or lost at least 4 months before the date of implantation
* Adequate bone quantity at the implant site to permit the insertion of a Straumann Standard or Standard Plus 4.1 mm diameter implant at least 8 mm in length without the use of concurrent bone augmentation techniques, i.e. Implant insertion sites must have sufficient bone height such that the implant will not encroach on vital structures and sufficient width that a minimum of 1 mm lingual and buccal bone will remain
* Patients must have signed the informed consent form. They must be committed to the study. If the treating clinicians doubt that the patient is willing or will be able to attend all study follow-up visits then the patient should not be admitted to the study

Exclusion Criteria:

* Patients with a history of systemic disease other than type 2 diabetes mellitus that may preclude dental implant therapy (including cardiovascular, hepatic, renal, gastrointestinal, metabolic, neurologic, pulmonary, endocrine, autoimmune, or psychiatric disorders)
* Presence of conditions requiring chronic routine prophylactic use of antibiotics (e.g., bacterial endocarditis, cardiac valvular anomalies, prosthetic joint replacements)
* Diabetic retinopathy requiring imminent or planned surgical intervention
* Diabetic neuropathy of sufficient severity as to require treatment for control of symptoms
* Serum creatinine > 1.6 mg/dl
* AST (SGOT) or ALT (AGPT) > 2 times upper limit of normal laboratory range
* Hypertension, with or without medications, having a systolic pressure > 185mm Hg or diastolic pressure > 105mm Hg
* Patient has significant untreated oral infections or inflammatory lesions
* Medical conditions requiring prolonged use of steroids
* History of leukocyte dysfunction and deficiencies
* History of bleeding disorders
* Patients with history of renal failure
* Patients with metabolic bone disorders
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Use of any investigational drug or device within the 30 day period immediately prior to implant surgery on study day 0
* Patients who smoke >10 cigarettes per day or cigar equivalents, or who chew tobacco
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, unreliability

Local Factors:

* Signs of oral inflammation, such as untreated periodontitis around the teeth or erosive lichen planus in the non-tooth associated areas
* History of head/neck irradiation therapy
* Presence of bone defects in the jaw preventing implant placement
* Unhealed extraction sites (less than 4 months post extraction of teeth in intended sites)
* Bone surgery (bone grafts, guided tissue regeneration technique for bone enhancement) less than 6 months prior to implant placement
* Patients requiring bone grafting at the surgical sites at the time of surgery
* Severe teeth grinding or clenching habits
* Persistent intraoral infection
* Lack of sufficient stability of the implant at surgery to allow for proper healing.
* Patients with inadequate oral hygiene or unmotivated for adequate home care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: thomas w oates, dmd, phd, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dental Implant: standard SLA surface and chemically-modified surface implant
Period: Overall Study
Arm/Group | Dental Implant
Started | 24
Completed | 18
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- Dental Implant: standard SLA surface and chemically modified surface
  dental implant : standard SLA surface and modified dental implant : chemically modified surface
Arm/Group | Dental Implant
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Implant Stability Quotient (ISQ)
Description: resonance frequency analysis employed to determine implant stability quotient on a 1-100 point scale with 100 representing the greatest stability.
Time Frame: 4 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- SLA Minimum ISQ HbA1c<9.5: standard SLA surface
  dental implant : standard SLA surface
- Modified SLA Minimum ISQ HbA1c<9.5: chemically modified surface
  modified dental implant : chemically modified surface
Arm/Group | SLA Minimum ISQ HbA1c<9.5 | Modified SLA Minimum ISQ HbA1c<9.5
Number analyzed (Participants) | 24 | 24
units on a scale | 61.9 (5.6) | 61.3 (3.2)

2. Secondary Outcome: Clinical Success of Implants
Time Frame: 1 year
Population: Data were not collected
Groups:
- Clinical Success of Implants: Successful outcome of implant after one year
Arm/Group | Clinical Success of Implants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Dental Implant: standard SLA surface
  dental implant : standard SLA surface
- Modified Dental Implant: chemically modified surface
  modified dental implant : chemically modified surface
Arm/Group | Dental Implant | Modified Dental Implant
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No